CLINICAL TRIAL: NCT01745744
Title: Clinical Trial Phase I / II, Multicentre, Open, Randomized Study of the Use of Mesenchymal Stem Cells From Adipose Tissue (CeTMAd) as Cell Regeneration Therapy in Critical Chronic Ischemic Syndrome of Lower Limb in Nondiabetic Patients.
Brief Title: Application of Cell Regeneration Therapy With Mesenchymal Stem Cells From Adipose Tissue in Critical Chronic Ischemic Syndrome of Lower Limbs (CLI) in Nondiabetic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CeTMAd/ICC/2009; 2009-013554-32 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): - Infusion of mesenchymal stem cells from adipose tissue: 0.5x106 cells / kg of patient weight.
  Interventions: Other: Mesenchymal stem cells from adipose tissue
- High dose (Experimental): - Infusion of mesenchymal stem cells from adipose tissue: 1x106 cells / kg of patient weight.
  Interventions: Other: Mesenchymal stem cells from adipose tissue
- Control (No Intervention): Conventional treatment

INTERVENTIONS:
Other: Mesenchymal stem cells from adipose tissue — - Infusion of mesenchymal stem cells from adipose tissue administered intraarterially: 0.5x106 cells / kg of patient weight and 1x106 cells / kg of patient weight.
  Arms: High dose; Low dose

SUMMARY:
Clinical trial phase I / II, prospective, multicenter, open, randomized, parallel-groups controlled by two levels of dose to assess the safety and feasibility of the infusion of mesenchymal stem cells from adipose tissue administered intra-arterially in nondiabetic patients with chronic ischemia of lower limbs (CLI) and no possibility of revascularization.

DETAILED DESCRIPTION:
A prospective, multicenter, open, randomized, parallel-group controlled study for two levels of dose.

The study population will consist of 30 non-diabetic patients with critical chronic ischemia in at least one of the lower limbs (CLI) and without possibility of revascularization, from whom results can clinically be evaluable, of whom, 20 patients will be included in the experimental group (10 for each dose level) and 10 in the control group.

In each of the two dose levels to be used in the study, 15 patients will be included, who will be randomized to the experimental group or the control group according to a distribution 2:1 (2 patients in the experimental group and 1 in control group), thus at each dose level, we will have 10 patients in the experimental group (treated with mesenchymal cells of adipose tissue) and 5 patients in the control group (conventional treatment, including the use of prostaglandins per protocol).

Patients who are randomized to experimental treatment Group with CeTMAd may receive one of the following dose levels:

* 0.5x106 cells / kg of patient weight
* 1x106 cells / kg of patient weight

The recruitment will be done with escalating doses, starting at the lower dose. To switch to the higher dose will require a favorable opinion of the Ethics Committee of the H. Universitario Virgen Macarena to evaluate the clinical status of patients and therapeutic safety and study procedures.

Patients who are randomized to the treatment control group will continue with conventional treatment which they were performing at the time of inclusion in the study (including the use of prostaglandins as protocol).

STUDY OBJECTIVE: To evaluate the safety and feasibility of regenerative treatment with mesenchymal stem cells from adipose tissue (CeTMAd), administered intraarterial in nondiabetic patients with chronic critical ischemia of at least one lower limb without possibilities of revascularization or alternative therapies. We will analyze the complications from regenerative therapy and / or study procedures.

* Main objectives:

  1. Security: It will be studied the possible complications due to the procedure in the first 24 hours of administration of CeTMAd, 1 month, 3 months, 6 months, 9 months and 12 months.
  2. Efficiency: It will be studied the generation of new vessels (vasculogenesis) and enhancement of collateral circulation (angiogenesis / arteriogenesis).
* Secondary objectives:

It will be studied the evolution of ankle brachial index, transcutaneous oxygen pressure, degree of Rutherford-Becker, ulcer size, calf perimeter, the score of pain and intermittent claudication (walking test).

Duration of the clinical trial: From the infusion to the patient of the Mesenchymal Stem Cells from Adipose Tissue to the end of the monitoring, there will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 18 and ≤ 89 years.
* Nondiabetic.
* Infrapopliteal atherosclerotic vascular disease of severe grade with either severe claudication or Rutherford-Becker grade II-III-IV, of at least one lower limb. It is defined critical ischemia of the lower limb as persistent/recurrent pain requiring analgesia and / or non-healing present ulcers > 4 weeks, with no evidence of improvement with conventional therapies and / or walking test (stress test) between 1-6 minutes in two exercise tests separated by at least 2 weeks and / or ankle-brachial index at rest <0.8.
* Inability of surgical or endovascular revascularization as recommended by the TransAtlantic InterSociety Consensus (TASC).
* Failure in the revascularization surgery performed at least 30 days before, with persistence or entry in critical ischemia phase.
* Life expectancy> 2 years.
* Not expected major amputation in the limb to treat in the next 12 months after inclusion.
* Normal biochemical parameters defined by:

  1. Leukocytes ≥ 3000
  2. Neutrophils ≥ 1500
  3. Platelets ≥ 100,000
  4. Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) ≤ 2.5 standard range institution
  5. Creatinine ≤ 2.5 mg / dl.
* Patients give their written informed consent to participate in the study.
* Women of childbearing potential must have negative results on a pregnancy test done at the time of inclusion in the study and agree to use a medically approved method of contraception for the duration of the study.

Exclusion Criteria:

* History of malignancy or hematologic disease (myeloproliferative disease, myelodysplastic syndrome or leukemia) in the last two years.
* Patients with uncontrolled hypertension (defined as blood pressure> 180/110 on more than one occasion).
* Severe heart failure (New York Heart Association class IV) or ejection fraction of the left ventricle less than 30%.
* Patients with malignant ventricular arrhythmias or unstable angina at the time of infusion.
* Diagnosis of deep vein thrombosis in the previous 3 months.
* Active infection or wet gangrene at day of infusion of Mesenchymal Stem Cells from Adipose Tissue.
* Concomitant therapy including hyperbaric oxygen. It is allowed the use of antiplatelet agents.
* Body mass index>40 kg/m2.
* Patients with a diagnosis of alcoholism at the time of inclusion.
* Untreated proliferative retinopathy.
* Concomitant disease that reduces life expectancy to less than a year.
* Predicted impossibility to obtain a biopsy providing 10 g of adipose tissue.
* human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
* Difficulty in monitoring.
* Stroke or myocardial infarction within the last 3 months.
* Anemia (hemoglobin <7.9 mg / dl).
* Leukopenia.
* Thrombocytopenia (<100,000 platelets / ul).
* Pregnant women or women of childbearing age who do not have adequate contraception.
* Patients who participated in a clinical trial within the last 3 months prior to inclusion in this clinical trial.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | 12 months.
  Number of adverse events and serious adverse events: 24h administration of CeTMAd, 1 month, 3 months, 6 months, 9 months and 12 months.

SECONDARY OUTCOMES:
Evolution of chronic critical ischemia | 1 month, 3 months, 6 months, 9 months and 12 months
  Parameters:Ankle brachial index, transcutaneous oxygen pressure, degree of Rutherford-Becker, larger ulcer size (as Texas classification), twin perimeter, score of pain and intermittent claudication (walking test).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael J. Ruiz-Salmerón, Principal Investigator — Hemodynamics Unit. Hospital Universitario Virgen Macarena.; Antonio de la Cuesta, Principal Investigator — Chronic Critical Ischemia Unit. San Lazaro Hospital.
Locations (2):
- Spain (2):
  - Hospital San Lazaro, Seville
  - University Hospital Virgen Macarena, Seville

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es